CLINICAL TRIAL: NCT05921760
Title: A Phase 1/2, Safety Lead-in and Dose Expansion, Open-label, Multicenter Trial Investigating the Safety, Tolerability, and Preliminary Activity of Ivosidenib in Combination With Nivolumab and Ipilimumab in Previously Treated Subjects With Nonresectable or Metastatic Cholangiocarcinoma With an IDH1 Mutation
Brief Title: Ivosidenib, Nivolumab, and Ipilimumab Combination in Previously Treated Subjects With Nonresectable or Metastatic IDH1 Mutant Cholangiocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study during the safety lead-in phase.
Sponsor: Servier Bio-Innovation LLC (Industry)
Collaborators: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL1-95031-006
Record Dates: First submitted 2023-04-21; First posted 2023-06-27 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: IDH1-mutant Cholangiocarcinoma
MeSH Terms: interventions — ivosidenib; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Lead-In Phase - Ivosidenib 500mg (Experimental)
  Interventions: Drug: Ivosidenib; Drug: Nivolumab; Drug: Ipilimumab
- Safety Lead-In Phase - Ivosidenib 250mg (Experimental)
  Interventions: Drug: Ivosidenib; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Ivosidenib — ivosidenib taken once daily
Drug: Nivolumab — Nivolumab taken by intravenous infusion
Drug: Ipilimumab — Ipilimumab taken by intravenous infusion

SUMMARY:
This is a Phase 1/2 study evaluating the safety, tolerability, and activity of ivosidenib in combination with immunotherapy in participants with nonresectable or metastatic cholangiocarcinoma. The study includes two phases: the safety lead-in phase to determine the recommended combination dose (RCD) of ivosidenib in combination with immunotherapy and the dose expansion phase to assess the efficacy of ivosidenib in combination with immunotherapy. Study treatment will be administered until participant experiences unacceptable toxicity, disease progression, or other discontinuation criteria are met.

This study was terminated by the sponsor before the expansion phase began and therefore participants were only involved in the safety lead-in phase.

ELIGIBILITY:
Inclusion Criteria:

* Male of female participant age ≥ 18 years old
* Have documented IDH1 gene-mutated disease based on local testing procedure (R132C/L/G/H/S mutations variants tested)
* Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1
* Has a histopathological diagnosis consistent with nonresectable or metastatic cholangiocarcinoma and are not eligible for curative resection, transplantation, or ablative therapies
* Participants must have at least one measurable lesion as defined by RECIST Version 1.1. Subjects who have received prior local therapy (including but not limited to embolization, chemoembolization, radiofrequency ablation, or radiation therapy) are eligible provided measurable disease falls outside of the treatment field or if within the field but has shown ≥ 20% growth in size post-treatment assessment.

Exclusion Criteria:

* Received prior treatment with an IDH inhibitor or prior treatment with an immune checkpoint inhibitor other than anti-PD1/L1
* Have active autoimmune disease or any condition requiring systemic treatment with either corticosteroids (> 10 mg daily of prednisone equivalents) or other immunosuppressive medications within 14 days of study treatment
* Participants who have not recovered from toxicity of previous anticancer therapy, including Grade ≥ 1 non-hematologic toxicity, according to the National Cancer Institute Common Terminology Criteria for Adverse Events v5.0, prior to the first IMP administration. Residual Grade ≤ 2 toxicity from chemotherapy (e.g., alopecia, neuropathy) may be allowed.
* Have known symptomatic brain metastases requiring steroids. Subjects with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study entry, have discontinued corticosteroid treatment for these metastases for at least 4 weeks, and have radiographically stable disease for at least 3 months prior to study entry. Note: Up to 10 mg per day of prednisone equivalent will be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - UCSF - Medical Center at Mission Bay, San Francisco, California
  - Ucsf Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
- UCLH, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/

REFERENCES:
- [Background] Kelley RK, Cleary JM, Sahai V, Baretti M, Bridgewater JA, Hua Z, Gliser C, Bian Y, Abou-Alfa GK. A phase 1/2, safety lead-in and dose expansion, open-label, multicenter trial investigating the safety, tolerability, and preliminary activity of ivosidenib in combination with nivolumab and ipilimumab in previously treated subjects with IDH1-mutated nonresectable or metastatic cholangiocarcinoma. J Clin Oncol. 2024 May 29;42(16_Supplement):TPS4197. doi: https://doi.org/10.1200/JCO.2024.42.16_suppl.TPS4197

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Started | 4 | 3
Completed | 0 | 0
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 3 | 2
Not completed — Sponsor Terminated the Study | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (20.61) | 49.3 (15.37) | 55.9 (18.12)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 2 | 2 | 4
  ≥ 65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  White | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 3 | 3 | 6
  Missing | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5
  United Kingdom | 0 | 2 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.80 (6.347) | 23.33 (2.114) | 25.31 (5.007)

OUTCOME MEASURES:

1. Primary Outcome: Safety Lead-In Phase: Number of Dose Limiting Toxicities (DLTs) Associated With Study Drug Regimen, During the First 2 Cycles of Treatment
Description: Occurring during the safety lead-in phase
Time Frame: Through the end of Cycle 2, day 42 (Cycle 1 and 2 are each 21 days)
Measure: Number; unit: DLT events
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 4 | 3
DLT events | 0 | 1

2. Primary Outcome: Safety Lead-In Phase: Number of Adverse Events (AEs)
Description: Occurring during the safety lead-in phase
Time Frame: Through study termination (approximately 1 year)
Measure: Number; unit: events
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 4 | 3
events | 71 | 27

3. Primary Outcome: Safety Lead-In Phase: Number of Participants With Adverse Events of Special Interests (AESIs)
Description: Occurring during the safety lead-in phase
Time Frame: Through study termination (approximately 1 year)
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

4. Primary Outcome: Safety Lead-In Phase: Number of Serious Adverse Events (SAEs)
Description: Occurring during the safety lead-in phase
Time Frame: Through study termination (approximately 1 year)
Measure: Number; unit: events
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 4 | 3
events | 3 | 2

5. Secondary Outcome: Safety Lead-In Phase: Area Under the Concentration-vs-time Curve (AUC) From 0 to Time of Last Measurable Concentration (AUC0-t)
Description: Occurring during the safety lead-in phase
Time Frame: Up to 3 years
Population: PK and PD samples were not analyzed due to the premature stop of the study and several dosing interruptions. The samples will not be analyzed in the future. Therefore, there is no parameter data available to be entered for this outcome measure.
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Safety Lead-In Phase: Plasma 2-hydroxyglutarate (2-HG) Concentration
Description: Occurring during the safety lead-in phase
Time Frame: up to 3 years
Population: as for outcome 5
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Safety Lead-In Phase: AUC Over 1 Dosing Interval at Steady State (AUCtau,ss)
Description: Occurring during the safety lead-in phase
Time Frame: Up to 3 years
Population: as for outcome 5
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Safety Lead-In Phase: Time to Maximum Concentration (Tmax)
Description: Occurring during the safety lead-in phase
Time Frame: Up to 3 years
Population: as for outcome 5
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Safety Lead-In Phase: Maximum Concentration (Cmax)
Description: Occurring during the safety lead-in phase
Time Frame: Up to 3 years
Population: as for outcome 5
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Safety Lead-In Phase: Trough Concentration (Ctrough)
Description: Occurring during the safety lead-in phase
Time Frame: Up to 3 years
Population: as for outcome 5
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Safety Lead-In Phase: Apparent Volume of Distribution (Vd/F)
Description: Occurring during the safety lead-in phase
Time Frame: Up to 3 years
Population: as for outcome 5
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Safety Lead-In Phase: Apparent Clearance (CL/F)
Description: Occurring during the safety lead-in phase
Time Frame: Up to 3 years
Population: as for outcome 5
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study termination (approximately 1 year)
Description: Adverse events were collected during participant visits.
Groups:
- Safety Lead-In Phase - Ivosidenib 500mg; Safety Lead-In Phase - Ivosidenib 250mg: First phase of the study.
  Ivosidenib: ivosidenib taken once daily
  Nivolumab: Nivolumab taken by intravenous infusion
  Ipilimumab: Ipilimumab taken by intravenous infusion
Arm/Group | Safety Lead-In Phase - Ivosidenib 500mg | Safety Lead-In Phase - Ivosidenib 250mg
All-Cause Mortality (participants affected / at risk) | 3/4 | 2/3
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Lead-In Phase - Ivosidenib 500mg (N=4) | Safety Lead-In Phase - Ivosidenib 250mg (N=3)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Lead-In Phase - Ivosidenib 500mg (N=4) | Safety Lead-In Phase - Ivosidenib 250mg (N=3)
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0
Malignant ascites (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 4 | 1
Pyrexia (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Candida infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Cardiac murmur (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Taste disorder (Nervous system disorders) | 2 | 0
Burning sensation (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT05921760/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT05921760/SAP_001.pdf